CLINICAL TRIAL: NCT01813435
Title: GLOBAL LEADERS: A Clinical Study Comparing Two Forms of Anti-platelet Therapy After Stent Implantation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ECRI bv (Industry)
Collaborators: Biosensors International (Other); AstraZeneca (Industry); The Medicines Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ECRI-12-001, 02EU11
Record Dates: First submitted 2013-02-12; First posted 2013-03-19 (Estimated); Results first posted 2019-07-05 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Coronary Artery Disease (CAD)
Keywords: CAD; ACS; All comers; DAPT; PCI
MeSH Terms: conditions — Coronary Artery Disease | interventions — Ticagrelor; Aspirin; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental treatment strategy (Experimental): All patients in the treatment group will receive acetylsalicylic acid (ASA) and ticagrelor for 1 month followed by 23 months of ticagrelor monotherapy.
  Dosage and frequency:
  Ticagrelor: 90 mg b.i.d. ASA: of 75mg qd (- ≤ 100 mg qd)
  Interventions: Drug: Ticagrelor; Drug: Acetylsalicylic Acid
- Reference treatment strategy (Active Comparator): Acute Coronary Syndrome (ACS) patients incl. unstable angina (UA) patients: ASA and Brilique(ticagrelor) for 12 months followed by 12 months of ASA monotherapy.
  Stable Coronary Artery Disease (CAD) patients: ASA and clopidogrel for 12 months followed by 12 months of ASA monotherapy.
  Dosage and frequency:
  Brilique(Ticagrelor): 90 mg b.i.d. ASA: of 75mg qd (- ≤ 100 mg qd) Clopidogrel: 75 mg qd
  Interventions: Drug: Ticagrelor; Drug: Acetylsalicylic Acid; Drug: Clopidogrel

INTERVENTIONS:
Drug: Ticagrelor — Comparison of 1 month of ticagrelor and aspirin followed by 23 months of ticagrelor monotherapy versus 12 months of standard dual anti platelet therapy (DAPT) followed by aspirin monotherapy.
  Other Names: Brilique
Drug: Acetylsalicylic Acid — Comparison of 1 month of ticagrelor and aspirin followed by 23 months of ticagrelor monotherapy versus 12 months of standard dual anti platelet therapy (DAPT) followed by aspirin monotherapy
  Other Names: Aspirin; B01AC06
Drug: Clopidogrel — Active Comparator: Reference treatment strategy Acute Coronary Syndrome (ACS) patients incl. unstable angina (UA) patients: ASA and Brilique(ticagrelor) for 12 months followed by 12 months of ASA monotherapy.
  Stable Coronary Artery Disease (CAD) patients: ASA and clopidogrel for 12 months followed by 12 months of ASA monotherapy
  Other Names: Plavix; B01AC04
  Arms: Reference treatment strategy

SUMMARY:
After a stent procedure, it is common practice to prescribe anti-platelet medication to prevent the blood from clotting. The main objective of this study is to determine if there is a better medication strategy to prevent blood from clotting and at the same time minimising the number of complications.

There are two medication strategies:

* Study group: Dual anti-platelet therapy (ticagrelor combined with aspirin) for 1 month, and then ticagrelor alone for another 23 months OR
* Control group: Standard treatment, being dual anti-platelet therapy (ticagrelor or clopidogrel combined with aspirin) for 12 months, and then aspirin alone indefinitely

DETAILED DESCRIPTION:
The study objective is to determine in all-comers patients undergoing percutaneous coronary intervention (PCI) under standardised treatment (including the BioMatrix family of drug-eluting stents and bivalirudin), whether treatment with 1 month of ticagrelor and aspirin followed by 23 months of ticagrelor monotherapy is superior with respect to the composite of all-cause mortality or non-fatal new Q-wave myocardial infarction (MI) compared to treatment with 12 months of standard dual anti platelet therapy (DAPT) followed by aspirin monotherapy.

The study design is an investigator-initiated, prospective randomised, multi-centre, multi-national, open-label trial to be conducted in approximately 60-80 interventional cardiology centres in Europe, North America, South America and Asia-Pacific. Patients will be randomised at a 1:1 ratio to study or reference treatment strategy.

Randomisation will occur at the time of the index procedure prior to PCI. Subjects will be stratified according to centre and according to the clinical presentation (Stable Coronary Artery Disease (CAD) vs. Acute Coronary Syndrome (ACS)).

All patients will be followed for a period of 2 years.

ELIGIBILITY:
Inclusion Criteria:

-"All comer" patients

1. Age ≥18 years;
2. Presence of one or more coronary artery stenoses of 50% or more in a native coronary artery or in a saphenous venous or arterial bypass conduit suitable for coronary stent implantation. The vessel should have a reference vessel diameter of at least 2.25 mm (no limitation on the number of treated lesions, vessels, or lesion length);
3. Able to provide informed consent and willing to participate in 2 year follow- up period.

Exclusion Criteria:

1. Known intolerance to aspirin, P2Y12 inhibitors, bivalirudin, stainless steel or biolimus;
2. Known intake of a strong CYP3A4 inhibitor (e.g., ketoconazole, clarithromycin, nefazodone, ritonavir, and atazanavir), as co-administration may lead to a substantial increase in exposure to ticagrelor;
3. Known moderate to severe hepatic impairment (alanine-aminotransferase ≥ 3 x ULN);
4. Planned surgery, including coronary artery bypass graft (CABG) as a staged procedure (hybrid) within 12 months of the index procedure, unless dual antiplatelet therapy is maintained throughout the peri-surgical period;
5. Need for chronic oral anti-coagulation therapy;
6. Active major bleeding or major surgery within the last 30 days;
7. Known history of intracranial haemorrhagic stroke or intra-cranial aneurysm;
8. Known stroke (any type) within the last 30 days;
9. Known pregnancy at time of randomisation;
10. Female who is breastfeeding at time of randomisation;
11. Currently participating in another trial and not yet at its primary endpoint.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15991 (Actual)
Dates: Start 2013-07-01 (Actual); Primary Completion 2015-11-09 (Actual); Study Completion 2018-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ernest Spitzer, MD, Study Director — European Cardiovascular Research Institute; Stephan Windecker, Prof. MD, Principal Investigator — Inselspital, University Hospital Bern, Switzerland
Locations (130):
- Australia (3):
  - Research centre Brisbane, 6101, Brisbane
  - Research centre Melbourne, 6104, Melbourne
  - Research centre Melbourne, 6105, Melbourne
- Austria (5):
  - Research centre Graz, 4305, Graz
  - Rsearch centre Innsbruck, 4303, Innsbruck
  - Research centre Linz, 4304, Linz
  - Research centre Vienna, 4301, Vienna
  - Research centre Vienna, 4302, Vienna
- Belgium (6):
  - Research centre Aalst, 3201, Aalst
  - Research centre Aalst, 3206, Aalst
  - Research centre Bonheiden, 3204, Bonheiden
  - Research centre Charleroi, 3202, Charleroi
  - Research centre Genk, 3205, Genk
  - Research centre Hasselt, 3203, Hasselt
- Brazil (5):
  - Research centre Rio de Janeiro, 5503, Rio de Janeiro
  - Research centre Rio de Janeiro, 5504, Rio de Janeiro
  - Research centre Sao Paulo, 5501, São Paulo
  - Research centre Sao Paulo, 5502, São Paulo
  - Research centre Uberlândia, 5505, Uberlândia
- Bulgaria (8):
  - Research centre Burgas, 9902, Burgas
  - Research centre Plovdiv, 9905, Plovdiv
  - Research centre Sofia, 9901, Sofia
  - Research centre Sofia, 9903, Sofia
  - Research centre Sofia, 9904, Sofia
  - Research centre Sofia, 9907, Sofia
  - Research centre Sofia, 9908, Sofia
  - Research centre Varna, 9906, Varna
- Canada (2):
  - Research centre Newmarket, 1003, Newmarket
  - Research centre Quebec, 1001, Québec
- Denmark (2):
  - Research centre Copenhagen, 4501, Copenhagen
  - Research centre Roskilde, 4503, Roskilde
- France (13):
  - Research centre Aix en Provence, 3311, Aix-en-Provence
  - Research centre Caen, 3308, Caen
  - Research centre Caen, 3309, Caen
  - Research centre Clermont-Ferrand, 3303, Clermont-Ferrand
  - Research centre Dijon, 3313, Dijon
  - Research centre Grenoble, 3312, Grenoble
  - Research centre Lyon, 3316, Lyon
  - Research centre Nancy, 3314, Nancy
  - Research centre Paris, 3301, Paris
  - Research centre Paris, 3305, Paris
  - Research centre Rouen, 3307, Rouen
  - Research centre Saint Etienne, 3310, Saint-Etienne
  - Research centre Toulouse, 3302, Toulouse
- Germany (17):
  - Research centre Bad Krozingen, 4904, Bad Krozingen
  - Research centre Bad Nauheim, 4902, Bad Nauheim
  - Research centre Berlin, 4918, Berlin
  - Research centre Bonn, 4911, Bonn
  - Research centre Dresden, 4908, Dresden
  - Research centre Essen, 4903, Essen
  - Research centre Fulda, 4905, Fulda
  - Research centre Giessen 4901, Giessen
  - Research centre Göttingen, 4907, Göttingen
  - Research centre Landshut, 4909, Landshut
  - Research centre Lubeck, 4917, Lübeck
  - Research centre Mainz, 4910, Mainz
  - Research centre Mannheim, 4912, Mannheim
  - Research centre Mönchengladbach, 4915, Mönchengladbach
  - Research centre Neuss, 4916, Neuss
  - Research centre Tubingen, 4914, Tübingen
  - Research centre Villingen - Schwenningen, 4919, Villingen-Schwenningen
- Hungary (8):
  - Research centre Balatonfüred, 3608, Balatonfüred
  - Research centre Budapest, 3602, Budapest
  - Research centre Budapest, 3603, Budapest
  - Research centre Debrecen, 3607, Debrecen
  - Research centre Gyula, 3606, Gyula
  - Research centre Nyíregyháza, 3605, Nyíregyháza
  - Research centre Pécs, 3604, Pécs
  - Research centre szeged, 3601, Szeged
- Italy (6):
  - Research centre Arezzo, 3902, Arezzo
  - Research centre Brescia, 3912, Brescia
  - Research centre Ferrara, 3905, Ferrara
  - Research centre Milano, 3901, Milan
  - Research centre Pavia, 3903, Pavia
  - Research centre Terni, 3909, Terni
- Netherlands (9):
  - Research centre Alkmaar, 3106, Alkmaar
  - OLVG Research centre Amsterdam, 3104, Amsterdam
  - UMCG Groningen, 3108, Groningen
  - Research centre Leeuwarden, 3102, Leeuwarden
  - Research centre Nieuwegein, 3107, Nieuwegein
  - Research centre Nijmegen, 3105, Nijmegen
  - EMC Rotterdam, 3101, Rotterdam
  - Maasstad Rotterdam, 3103, Rotterdam
  - Research centre Tilburg, 3109, Tilburg
- Poland (7):
  - Research centre Chrzanow, 4802, Chrzanów
  - Research centre Dabrowa Gornicza, 4801, Dąbrowa Górnicza
  - Research centre Kedzierzyn-Kozle, 4805, Kędzierzyn-Koźle
  - Research centre Krakov, 4807, Krakow
  - Research centre Mielec, 4809, Mielec
  - Research centre Nysa, 4808, Nysa
  - Research centre Ustroń, 4803, Ustroń
- Portugal (4):
  - Research centre Gaia, 3501, Gaia
  - Research centre Lisbon, 3503, Lisbon
  - Research centre Lisbon, 3504, Lisbon
  - Research centre Lisbon, 3505, Lisbon
- Singapore (2):
  - Research centre Singapore, 6501, Singapore
  - Research centre Singapore, 6502, Singapore
- Spain (9):
  - Research centre Barcelona, 3401, Barcelona
  - Research centre Barcelona, 3403, Barcelona
  - Research centre Barcelona, 3405, Barcelona
  - Research centre Huelva, 3408, Huelva
  - Research centre Madrid 3410, Madrid
  - Research centre Madrid, 3402, Madrid
  - Research centre Madrid, 3407, Madrid
  - Research centre Madrid, 3409, Madrid
  - Research centre Vigo, 3404, Vigo
- Switzerland (6):
  - Research centre Bern, 4106, Bern
  - Research centre Bern, 4107, Bern
  - Research centre Geneva, 4101, Geneva
  - Research centre Lausanne, 4104, Lausanne
  - Research centre Liestal, 4108, Liestal
  - Research centre Lugano, 4105, Lugano
- United Kingdom (18):
  - Research centre Belfast, 4420, Belfast
  - Research Centre Belfast, 4423, Belfast
  - Research centre Blackburn, 4404, Blackburn
  - Research centre Blackpool, 4408, Blackpool
  - Research centre Bournemouth, 4418, Bournemouth
  - Research centre Brighton, 4405, Brighton
  - Research centre Cambridge, 4417, Cambridge
  - Research centre Cardiff, 4402, Cardiff
  - Research centre Glasgow, 4407, Glasgow
  - Research centre Leicester, 4421, Leicester
  - Research centre Liverpool, 4001, Liverpool
  - Research centre Manchester, 4403, Manchester
  - Research centre Manchester, 4406, Manchester
  - Research centre Newcastle, 4413, Newcastle
  - Research centre Rhyl, 4414, Rhyl
  - Research centre Southampton, 4415, Southampton
  - Research centre Stevenage, 4412, Stevenage
  - Research centre Wolverhampton, 4422, Wolverhampton

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Vranckx P, Valgimigli M, Juni P, Hamm C, Steg PG, Heg D, van Es GA, McFadden EP, Onuma Y, van Meijeren C, Chichareon P, Benit E, Mollmann H, Janssens L, Ferrario M, Moschovitis A, Zurakowski A, Dominici M, Van Geuns RJ, Huber K, Slagboom T, Serruys PW, Windecker S; GLOBAL LEADERS Investigators. Ticagrelor plus aspirin for 1 month, followed by ticagrelor monotherapy for 23 months vs aspirin plus clopidogrel or ticagrelor for 12 months, followed by aspirin monotherapy for 12 months after implantation of a drug-eluting stent: a multicentre, open-label, randomised superiority trial. Lancet. 2018 Sep 15;392(10151):940-949. doi: 10.1016/S0140-6736(18)31858-0. Epub 2018 Aug 27. PMID 30166073
- [Derived] Woelders ECI, Onuma Y, Ninomiya K, O'Leary N, Damman P, Peeters DAM, Hof AWJV', Valgimigli M, Vranckx P, Windecker S, Serruys PWJC, van Geuns RM. Parsimonious versus extensive bleeding score: can we simplify risk stratification after percutaneous coronary intervention and reduce bleeding events by de-escalation of the antiplatelet strategy? Open Heart. 2025 Jan 28;12(1):e003083. doi: 10.1136/openhrt-2024-003083. PMID 39875171
- [Derived] Ono M, Hara H, Kawashima H, Gao C, Wang R, Wykrzykowska JJ, Piek JJ, Garg S, Hamm C, Steg PG, Valgimigli M, Windecker S, Vranckx P, Onuma Y, Serruys PW. Ticagrelor monotherapy versus aspirin monotherapy at 12 months after percutaneous coronary intervention: a landmark analysis of the GLOBAL LEADERS trial. EuroIntervention. 2022 Aug 5;18(5):e377-e388. doi: 10.4244/EIJ-D-21-00870. PMID 35260381
- [Derived] Gragnano F, Zwahlen M, Vranckx P, Heg D, Schmidlin K, Hamm C, Steg PG, Gargiulo G, McFadden EP, Onuma Y, Chichareon P, Benit E, Mollmann H, Janssens L, Leonardi S, Zurakowski A, Arrivi A, Van Geuns RJ, Huber K, Slagboom T, Calabro P, Serruys PW, Juni P, Valgimigli M, Windecker S; GLOBAL LEADERS Investigators [Link]. Ticagrelor Monotherapy or Dual Antiplatelet Therapy After Drug-Eluting Stent Implantation: Per-Protocol Analysis of the GLOBAL LEADERS Trial. J Am Heart Assoc. 2022 May 17;11(10):e024291. doi: 10.1161/JAHA.121.024291. Epub 2022 Mar 1. PMID 35229616
- [Derived] Westra J, Eftekhari A, Renkens M, Mejia-Renteria H, Sejr-Hansen M, Stegehuis V, Holm NR, de Winter RJ, Piek JJ, Escaned J, Wykrzykowska JJ, Christiansen EH. Characterization of quantitative flow ratio and fractional flow reserve discordance using doppler flow and clinical follow-up. Int J Cardiovasc Imaging. 2022 Jun;38(6):1181-1190. doi: 10.1007/s10554-022-02522-1. Epub 2022 Jan 18. PMID 35041147
- [Derived] Vranckx P, Valgimigli M, Odutayo A, Serruys PW, Hamm C, Steg PG, Heg D, Mc Fadden EP, Onuma Y, Benit E, Janssens L, Diletti R, Ferrario M, Huber K, Raber L, Windecker S, Juni P; GLOBAL LEADERS Investigators. Efficacy and Safety of Ticagrelor Monotherapy by Clinical Presentation: Pre-Specified Analysis of the GLOBAL LEADERS Trial. J Am Heart Assoc. 2021 Sep 21;10(18):e015560. doi: 10.1161/JAHA.119.015560. Epub 2021 Sep 17. PMID 34533034
- [Derived] Gao C, Tomaniak M, Takahashi K, Kawashima H, Wang R, Hara H, Ono M, Montalescot G, Garg S, Haude M, Slagboom T, Vranckx P, Valgimigli M, Windecker S, van Geuns RJ, Hamm C, Steg PG, Onuma Y, Angiolillo DJ, Serruys PW. Ticagrelor monotherapy in patients with concomitant diabetes mellitus and chronic kidney disease: a post hoc analysis of the GLOBAL LEADERS trial. Cardiovasc Diabetol. 2020 Oct 16;19(1):179. doi: 10.1186/s12933-020-01153-x. PMID 33066794
- [Derived] Kawashima H, Tomaniak M, Ono M, Wang R, Hara H, Gao C, Takahashi K, Sharif F, Thury A, Suryapranata H, Walsh S, Cotton J, Carrie D, Sabate M, Steinwender C, Leibundgut G, Wykrzykowska J, de Winter RJ, Garg S, Hamm C, Steg PG, Juni P, Vranckx P, Valgimigli M, Windecker S, Onuma Y, Serruys PW. Safety and Efficacy of 1-Month Dual Antiplatelet Therapy (Ticagrelor + Aspirin) Followed by 23-Month Ticagrelor Monotherapy in Patients Undergoing Staged Percutaneous Coronary Intervention (A Sub-Study from GLOBAL LEADERS). Am J Cardiol. 2021 Jan 1;138:1-10. doi: 10.1016/j.amjcard.2020.09.057. Epub 2020 Oct 13. PMID 33065080
- [Derived] Gao C, Takahashi K, Garg S, Hara H, Wang R, Kawashima H, Ono M, Montalescot G, Haude M, Slagboom T, Vranckx P, Valgimigli M, Windecker S, Hamm C, Steg PG, Storey R, van Geuns RJ, Tao L, Onuma Y, Serruys PW. Regional variation in patients and outcomes in the GLOBAL LEADERS trial. Int J Cardiol. 2021 Feb 1;324:30-37. doi: 10.1016/j.ijcard.2020.09.039. Epub 2020 Sep 15. PMID 32941872
- [Derived] Hara H, Takahashi K, Kogame N, Tomaniak M, Kerkmeijer LSM, Ono M, Kawashima H, Wang R, Gao C, Wykrzykowska JJ, de Winter RJ, Neumann FJ, Plante S, Lemos Neto PA, Garg S, Juni P, Vranckx P, Windecker S, Valgimigli M, Hamm C, Steg PG, Onuma Y, Serruys PW. Impact of Bleeding and Myocardial Infarction on Mortality in All-Comer Patients Undergoing Percutaneous Coronary Intervention. Circ Cardiovasc Interv. 2020 Sep;13(9):e009177. doi: 10.1161/CIRCINTERVENTIONS.120.009177. Epub 2020 Aug 25. PMID 32838554
- [Derived] Hara H, van Klaveren D, Takahashi K, Kogame N, Chichareon P, Modolo R, Tomaniak M, Ono M, Kawashima H, Wang R, Gao C, Niethammer M, Fontos G, Angioi M, Ribeiro VG, Barbato E, Leandro S, Hamm C, Valgimigli M, Windecker S, Juni P, Steg PG, Verbeeck J, Tijssen JGP, Sharif F, Onuma Y, Serruys PW; GLOBAL LEADERS Trial Investigators. Comparative Methodological Assessment of the Randomized GLOBAL LEADERS Trial Using Total Ischemic and Bleeding Events. Circ Cardiovasc Qual Outcomes. 2020 Aug;13(8):e006660. doi: 10.1161/CIRCOUTCOMES.120.006660. Epub 2020 Jul 30. PMID 32762446
- [Derived] Ono M, Chichareon P, Tomaniak M, Kawashima H, Takahashi K, Kogame N, Modolo R, Hara H, Gao C, Wang R, Walsh S, Suryapranata H, da Silva PC, Cotton J, Koning R, Akin I, Rensing BJWM, Garg S, Wykrzykowska JJ, Piek JJ, Juni P, Hamm C, Steg PG, Valgimigli M, Windecker S, Storey RF, Onuma Y, Vranckx P, Serruys PW. The association of body mass index with long-term clinical outcomes after ticagrelor monotherapy following abbreviated dual antiplatelet therapy in patients undergoing percutaneous coronary intervention: a prespecified sub-analysis of the GLOBAL LEADERS Trial. Clin Res Cardiol. 2020 Sep;109(9):1125-1139. doi: 10.1007/s00392-020-01604-1. Epub 2020 Jan 31. PMID 32006156
- [Derived] Tomaniak M, Chichareon P, Klimczak-Tomaniak D, Takahashi K, Kogame N, Modolo R, Wang R, Ono M, Hara H, Gao C, Kawashima H, Rademaker-Havinga T, Garg S, Curzen N, Haude M, Kochman J, Gori T, Montalescot G, Angiolillo DJ, Capodanno D, Storey RF, Hamm C, Vranckx P, Valgimigli M, Windecker S, Onuma Y, Serruys PW, Anderson R. Impact of renal function on clinical outcomes after PCI in ACS and stable CAD patients treated with ticagrelor: a prespecified analysis of the GLOBAL LEADERS randomized clinical trial. Clin Res Cardiol. 2020 Jul;109(7):930-943. doi: 10.1007/s00392-019-01586-9. Epub 2020 Jan 10. PMID 31925529
- [Derived] Tomaniak M, Chichareon P, Takahashi K, Kogame N, Modolo R, Chang CC, Spitzer E, Neumann FJ, Plante S, Hernandez Antolin R, Jambrik Z, Gelev V, Brunel P, Konteva M, Beygui F, Morelle JF, Filipiak KJ, van Geuns RJ, Soliman O, Tijssen J, Rademaker-Havinga T, Storey RF, Hamm C, Steg PG, Windecker S, Onuma Y, Valgimigli M, Serruys PW; GLOBAL LEADERS Study Investigators. Impact of chronic obstructive pulmonary disease and dyspnoea on clinical outcomes in ticagrelor treated patients undergoing percutaneous coronary intervention in the randomized GLOBAL LEADERS trial. Eur Heart J Cardiovasc Pharmacother. 2020 Jul 1;6(4):222-230. doi: 10.1093/ehjcvp/pvz052. PMID 31876907
- [Derived] Tomaniak M, Chichareon P, Modolo R, Takahashi K, Chang CC, Kogame N, Spitzer E, Buszman PE, van Geuns RM, Valkov V, Steinwender C, Geisler T, Prokopczuk J, Sabate M, Zmudka K, Rademaker-Havinga T, Tijssen JGP, Juni P, Hamm C, Steg PG, Onuma Y, Vranckx P, Valgimigli M, Windecker S, Baber U, Anderson R, Dominici M, Serruys PW. Ticagrelor monotherapy beyond one month after PCI in ACS or stable CAD in elderly patients: a pre-specified analysis of the GLOBAL LEADERS trial. EuroIntervention. 2020 Apr 3;15(18):e1605-e1614. doi: 10.4244/EIJ-D-19-00699. PMID 31845894
- [Derived] Chichareon P, Modolo R, Kerkmeijer L, Tomaniak M, Kogame N, Takahashi K, Chang CC, Komiyama H, Moccetti T, Talwar S, Colombo A, Maillard L, Barlis P, Wykrzykowska J, Piek JJ, Garg S, Hamm C, Steg PG, Juni P, Valgimigli M, Windecker S, Onuma Y, Mehran R, Serruys PW. Association of Sex With Outcomes in Patients Undergoing Percutaneous Coronary Intervention: A Subgroup Analysis of the GLOBAL LEADERS Randomized Clinical Trial. JAMA Cardiol. 2020 Jan 1;5(1):21-29. doi: 10.1001/jamacardio.2019.4296. PMID 31693078
- [Derived] Takahashi K, Serruys PW, Chichareon P, Chang CC, Tomaniak M, Modolo R, Kogame N, Magro M, Chowdhary S, Eitel I, Zweiker R, Ong P, Ottesen MM, Tijssen JGP, Wykrzykowska JJ, de Winter RJ, Garg S, Stoll HP, Hamm C, Steg PG, Onuma Y, Valgimigli M, Vranckx P, Carrie D, Windecker S. Efficacy and Safety of Ticagrelor Monotherapy in Patients Undergoing Multivessel PCI. J Am Coll Cardiol. 2019 Oct 22;74(16):2015-2027. doi: 10.1016/j.jacc.2019.08.997. PMID 31623758
- [Derived] Tomaniak M, Chichareon P, Onuma Y, Deliargyris EN, Takahashi K, Kogame N, Modolo R, Chang CC, Rademaker-Havinga T, Storey RF, Dangas GD, Bhatt DL, Angiolillo DJ, Hamm C, Valgimigli M, Windecker S, Steg PG, Vranckx P, Serruys PW; GLOBAL LEADERS Trial Investigators. Benefit and Risks of Aspirin in Addition to Ticagrelor in Acute Coronary Syndromes: A Post Hoc Analysis of the Randomized GLOBAL LEADERS Trial. JAMA Cardiol. 2019 Nov 1;4(11):1092-1101. doi: 10.1001/jamacardio.2019.3355. PMID 31557763
- [Derived] Serruys PW, Tomaniak M, Chichareon P, Modolo R, Kogame N, Takahashi K, Chang CC, Spitzer E, Walsh SJ, Adlam D, Hildick-Smith D, Edes I, van de Harst P, Krackhardt F, Tijssen JGP, Rademaker-Havinga T, Garg S, Steg PG, Hamm C, Juni P, Vranckx P, Onuma Y, Verheugt FWA. Patient-oriented composite endpoints and net adverse clinical events with ticagrelor monotherapy following percutaneous coronary intervention: insights from the randomised GLOBAL LEADERS trial. EuroIntervention. 2019 Dec 20;15(12):e1090-e1098. doi: 10.4244/EIJ-D-19-00202. PMID 30888959
- [Derived] Leonardi S, Franzone A, Piccolo R, McFadden E, Vranckx P, Serruys P, Benit E, Liebetrau C, Janssens L, Ferrario M, Zurakowski A, van Geuns RJ, Dominici M, Huber K, Slagboom T, Buszman P, Bolognese L, Tumscitz C, Bryniarski K, Aminian A, Vrolix M, Petrov I, Garg S, Naber C, Prokopczuk J, Hamm C, Steg G, Heg D, Juni P, Windecker S, Valgimigli M. Rationale and design of a prospective substudy of clinical endpoint adjudication processes within an investigator-reported randomised controlled trial in patients with coronary artery disease: the GLOBAL LEADERS Adjudication Sub-StudY (GLASSY). BMJ Open. 2019 Mar 9;9(3):e026053. doi: 10.1136/bmjopen-2018-026053. PMID 30852547
- See also: Pubmed Identifier 30166073 — http://dx.doi.org/10.1016/S0140-6736(18)31858-0

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 12 participants of the experimental group withdrew consent or objected to use further use of data
  11 participants of the reference group withdrew consent or objected to use further use of data
Groups:
- Experimental Treatment Strategy: All patients in the treatment group will receive acetylsalicylic acid (ASA) and ticagrelor for 1 month followed by 23 months of ticagrelor monotherapy.
  Dosage and frequency:
  Ticagrelor: 90 mg b.i.d. ASA: of 75mg qd (- ≤ 100 mg qd)
  Ticagrelor: Comparison of 1 month of ticagrelor and aspirin followed by 23 months of ticagrelor monotherapy versus 12 months of standard dual anti platelet therapy (DAPT) followed by aspirin monotherapy.
  Acetylsalicylic Acid: Comparison of 1 month of ticagrelor and aspirin followed by 23 months of ticagrelor monotherapy versus 12 months of standard dual anti platelet therapy (DAPT) followed by aspirin monotherapy
- Reference Treatment Strategy: Acute Coronary Syndrome (ACS) patients incl. unstable angina (UA) patients: ASA and Brilique(ticagrelor) for 12 months followed by 12 months of ASA monotherapy.
  Stable Coronary Artery Disease (CAD) patients: ASA and clopidogrel for 12 months followed by 12 months of ASA monotherapy.
  Dosage and frequency:
  Brilique(Ticagrelor): 90 mg b.i.d. ASA: of 75mg qd (- ≤ 100 mg qd) Clopidogrel: 75 mg qd
  Ticagrelor: Comparison of 1 month of ticagrelor and aspirin followed by 23 months of ticagrelor monotherapy versus 12 months of standard dual anti platelet therapy (DAPT) followed by aspirin monotherapy.
  Acetylsalicylic Acid: Comparison of 1 month of ticagrelor and aspirin followed by 23 months of ticagrelor monotherapy versus 12 months of standard dual anti platelet therapy (DAPT) followed by aspirin monotherapy
  Clopidogrel: Active Comparator: Reference treatment strategy Acute Coronary Syndrome (ACS) patients incl. unstable angina (UA) patients: ASA and Brilique(ticagrelor) for
Period: Overall Study
Arm/Group | Experimental Treatment Strategy | Reference Treatment Strategy
Started | 7980 (12 participants withdrew consent or objected to use further use of data) | 7988 (11 participants withdrew consent or objected to use further use of data)
Completed | 5810 | 6981
Not Completed | 2170 | 1007
Not completed — did not finish experimental regimen | 1902 | 770
Not completed — Lost to Follow-up | 268 | 237

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental Treatment Strategy | Reference Treatment Strategy | Total
Number analyzed (Participants) | 7980 | 7988 | 15968
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3949 | 3928 | 7877
  >=65 years | 4031 | 4060 | 8091
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.5 (10.3) | 64.6 (10.3) | 64.6 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: these are the numbers analysed for primary endpoint.
  Participants
    Female | 1865 | 1849 | 3714
    Male | 6115 | 6139 | 12254
Region of Enrollment [Number; unit: participants]
  Singapore | 71 | 71 | 142
  Hungary | 264 | 263 | 527
  United Kingdom | 854 | 859 | 1713
  Portugal | 56 | 57 | 113
  Switzerland | 352 | 353 | 705
  Spain | 475 | 476 | 951
  Canada | 84 | 86 | 170
  Austria | 335 | 337 | 672
  Netherlands | 579 | 580 | 1159
  Belgium | 1094 | 1091 | 2185
  Brazil | 126 | 122 | 248
  Denmark | 66 | 65 | 131
  Poland | 768 | 764 | 1532
  Italy | 790 | 788 | 1578
  Australia | 41 | 42 | 83
  Bulgaria | 470 | 473 | 943
  France | 426 | 423 | 849
  Germany | 1129 | 1138 | 2267

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Composite of All-cause Mortality or Non-fatal New Q-wave Myocardial Infarction (MI)
Description: Number of Participants with a composite of all-cause mortality or non-fatal new Q-wave MI up to 2 years post randomisation.
Time Frame: 2 year
Population: Shown are the first event per event type for each patient only. Multiple events of the same type within the same patient are disregarded. Data were censored 730 days after index percutaneous coronary intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Treatment Strategy | Reference Treatment Strategy
Number analyzed (Participants) | 7980 | 7988
Participants | 304 | 349

2. Secondary Outcome: Number of Participants With All-cause Mortality
Time Frame: 2-year
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Treatment Strategy | Reference Treatment Strategy
Number analyzed (Participants) | 7980 | 7988
Participants | 224 | 253

3. Secondary Outcome: Number of Participants With Myocardial Infarction
Time Frame: 2 year
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Treatment Strategy | Reference Treatment Strategy
Number analyzed (Participants) | 7980 | 7988
Participants | 248 | 250

4. Secondary Outcome: Number of Participants With New Q-wave Myocardial Infarction
Time Frame: 2-year
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Treatment Strategy | Reference Treatment Strategy
Number analyzed (Participants) | 7980 | 7988
Participants | 83 | 103

5. Secondary Outcome: Number of Participants With a Composite of All-cause Mortality, Stroke, or New Q-wave Myocardial Infarction
Description: shown are the first event per event type for each patient only. Multiple events of the same type within the same patient are disregarded
Time Frame: 2-year
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Treatment Strategy | Reference Treatment Strategy
Number analyzed (Participants) | 7980 | 7988
Participants | 362 | 416

6. Secondary Outcome: Number of Participants With a Stroke
Time Frame: 2 year
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Treatment Strategy | Reference Treatment Strategy
Number analyzed (Participants) | 7980 | 7988
Participants | 80 | 82

7. Secondary Outcome: Number of Participants With a Myocardial Revascularisation
Time Frame: 2 year
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Treatment Strategy | Reference Treatment Strategy
Number analyzed (Participants) | 7980 | 7988
Participants | 739 | 793

8. Secondary Outcome: Number of Participants With a Definite Stent Thrombosis
Time Frame: 2 year
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Treatment Strategy | Reference Treatment Strategy
Number analyzed (Participants) | 7980 | 7988
Participants | 64 | 64

9. Secondary Outcome: Number of Participants With a Bleeding Academic Research Consortium (BARC) 3 or 5 Bleeding
Description: BARC definition. We only considered BARC 3 or 5 for this secondary safety endpoint.
  Type 3: Clinical, laboratory, and/or imaging evidence of bleeding with:
  * Type 3a:
    * Overt bleeding + Hb drop of 3 to < 5 g/dL (provided Hb drop is related to bleed)
    * Any transfusion with overt bleeding
  * Type 3b:
    * Overt bleeding + Hb drop ≥5 g/dL (provided Hb drop is related to bleed)
    * Cardiac tamponade
    * Bleeding requiring surgical intervention (excluding dental/nasal/skin/haemorrhoid)
    * Bleeding requiring intravenous vasoactive agents
  * Type 3c:
    * Intracranial haemorrhage (does not include microbleeds or haemorrhagic transformation, does include intraspinal)
    * Subcategories confirmed by autopsy or imaging or lumbar puncture
    * Intraocular bleed compromising vision. Type 5: Fatal bleeding
    * Type 5a:
      • Probable fatal bleeding; no autopsy or imaging confirmation but clinically suspicious
    * Type 5b:
      * Definite fatal bleeding; overt bleeding or autopsy or imaging confirmation
Time Frame: 2 year
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Treatment Strategy | Reference Treatment Strategy
Number analyzed (Participants) | 7980 | 7988
Participants | 163 | 169

ADVERSE EVENTS:
Time Frame: monitored for 2 years
Arm/Group | Experimental Treatment Strategy | Reference Treatment Strategy
All-Cause Mortality (participants affected / at risk) | 224/7980 | 253/7988
Serious Adverse Events (participants affected / at risk) | 1459/7980 | 1543/7988
Other Adverse Events (participants affected / at risk) | 0/7980 | 0/7988
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental Treatment Strategy (N=7980) | Reference Treatment Strategy (N=7988)
new Q-wave MI (Cardiac disorders) | 83 | 103
MI (Cardiac disorders) | 248 | 250
stroke (Vascular disorders) | 162 | 164
revascularisation (Vascular disorders) | 739 | 793
definite stent thrombosis (Vascular disorders) | 64 | 64
BARC 3 or 5 bleeding (Vascular disorders) | 163 | 169

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes